CLINICAL TRIAL: NCT05160051
Title: 68Ga-FAPI-46 PET for Imaging of FAP Expressing Cancer: A Single-center Prospective Interventional Single-arm Clinical Trial
Brief Title: 68Ga-FAPI-46 PET for Imaging of FAP Expressing Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital, Essen (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: FAPI-PET Trial
Record Dates: First submitted 2021-10-12; First posted 2021-12-16 (Actual); Last update posted 2024-04-12 (Actual); Status verified 2024-04

CONDITIONS: Tumor, Solid
Keywords: radiotracer; PET scan; FAPI-46; 68Ga-radiotracer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Intervention Model Description: Single application of 68Ga-68-FAPI-46 PET/CT imaging to detect tumour tissue in patients with newly diagnosed or recurrent cancer
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 68Ga-FAPI-46 PET Scan (Experimental): A single-center prospective interventional single-arm clinical trial. All eligible subjects undergo FAPI-PET Scan
  Interventions: Diagnostic Test: 68Ga-FAPI-46 PET Scan

INTERVENTIONS:
Diagnostic Test: 68Ga-FAPI-46 PET Scan — 68Ga-FAPI-46 is a radiotracer that binds with high affinity to Fibroblast Activating Protein (FAP). FAP is physiologically expressed in many tissues during embryonic development, but in adults it is expressed only in the context of wound healing, fibrotic processes, and the stroma of many malignancies. Therefore, the study seeks to validate if 68Ga-FAPI-46 PET could be established as a diagnositc tool to detect solid tumors.

SUMMARY:
This study is to explore the safety and tolerability as well as diagnostic accuracy of 68Ga-FAPI-46 for different FAP-expressing tumor entities by PET.

This study does not offer any treatment for patients with FAP-expressing carcinomas; therefore, patients will be offered state of the art therapeutic options. Routine surgery will be performed within 8 weeks after 68Ga-FAPI-46 PET.

DETAILED DESCRIPTION:
Primary Endpoint:

Positive predictive value (PPV) on a per-region- and per-patient-basis of 68Ga-FAPI-46 PET for detection of histopathology-FAPpositive tumor lesions, confirmed by histopathology/biopsy (reached for ≥ 75%).

Secondary Endpoints:

1. Association between 68Ga-FAPI-46 PET uptake intensity and histopathologic FAP expression
2. Sensitivity and specificity of 68Ga-FAPI-46 PET on a per-patient and per-region-basis for detection of histopathology-FAPpositive tumor lesions confirmed by histopathology/biopsy (separate for regional, extra-regional and distant locations)
3. Detection rate of 68Ga-FAPI-46 PET versus previous standard imaging on a per-patient and per-region-basis for detection of tumor location, also stratified by tumor maker serum level
4. Sensitivity and specificity of 68Ga-FAPI-46 PET versus previous standard imaging on a per-patient and per-region-basis for detection of tumor lesions confirmed by combined histopathology/biopsy/follow-up imaging/clinical follow-up reference standard (separate for regional, extra-regional and distant locations)
5. Impact on management
6. Inter-reader reproducibility
7. Safety
8. Change in staging/prognostic groups

ELIGIBILITY:
Inclusion Criteria:

1. Proven or suspected tumor types: Breast, Colorectal, Endometrial, Esophageal, Glioma/GMB, Head and neck, Hepatocellular carcinoma, ,Lymphoma, Multiple Myeloma, Neuroendocrine, NSCLC (Non small cell lung cancer), Ovarian, Pancreatic, Prostate, Renal cell carcinoma, Sarcoma, SCLC (Small cell lung cancer), Semimoma, Thyroid, Unknown primary, Other
2. At initial staging or re-staging of disease
3. At least one detectable tumor lesion with any diameter >1 cm
4. Intended or performed surgery or biopsy of tumor within 8 weeks before or after enrollment
5. Age ≥18 years
6. Patient Eastern Cooperative Oncology Group (ECOG) performance status ≤2.
7. Women of child bearing potential (WOCBP), defined as all women physiologically capable of becoming pregnant, can only be included after a confirmed menstrual period and a negative highly sensitive urine or serum pregnancy test within 24 h before radiopharmaceutical application.

Exclusion Criteria:

1. Patient cannot give consent for the study
2. Patient cannot lie flat or tolerate 68Ga-FAPI-46 PET imaging
3. Prior external beam radiation therapy (EBRT) within 3 months of enrollment to tumor lesions intended for surgery or biopsy
4. Prior chemotherapy, immunotherapy, biologic or targeted oncologic therapy within 3 months of enrollment
5. Unwillingness or inability to comply with study and follow-up procedures
6. History of disease or condition that may critically interfere with participation in this study at the discretion of the investigators
7. Pregnant, lactating, or breast-feeding women
8. Women of child bearing potential (WOCBP), defined as all women physiologically capable of becoming pregnant, are not allowed to participate in this study, unless they are using highly effective methods of contraception during the interventional period. Highly effective contraception methods include:

   * True sexual abstinence: defined as refraining from heterosexual intercourse, when this is in line with the preferred and usual lifestyle of the patient. Periodic abstinence (e.g., calendar, ovulation, symptothermal, postovulation methods), declaration of abstinence for the duration of exposure to IMP, and withdrawal are not acceptable methods of contraception.
   * Vasectomised partner is a highly effective birth control method if the partner is the sole sexual partner of the study participant and the vasectomised partner has received medical assessment of the surgical success.
   * Bilateral tubal occlusion.
   * Combined (estrogen- and progestogen-containing) hormonal contraception associated with inhibition of ovulation:

     * oral
     * intravaginal
     * transdermal
   * Progestogen-only hormonal contraception associated with inhibition of ovulation:

     * oral
     * injectable
     * implantable
   * Placement of an intrauterine device (IUD) or intrauterine hormone-releasing system (IUS)
9. Post-menopausal women are allowed to participate in this study. Women are considered post-menopausal and not of child bearing potential if they have had 12 months of natural (spontaneous) amenorrhea with an appropriate clinical profile (e.g. age appropriate, history of vasomotor symptoms), or six months of spontaneous amenorrhea with serum folliclestimulating hormone (FSH) levels > 40mIU/mL or have had surgical bilateral oophorectomy or bilateral salpingectomy or hysterectomy or tubal ligation at least six weeks prior to screening. In the case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow up hormone level assessment is she considered not of child bearing potential
10. Sexually active males must use a condom during intercourse during the interventional period. A condom is required to be used also by vasectomized men in order to prevent delivery of the study compound via seminal fluid
11. QTcF >470 msec for females and QTcF >450 msec for males on screening electrocardiogram (ECG) or history of congenital long QT syndrome.
12. Known or expected hypersensitivity to 68Ga-68-FAPI-46 or any of the relevant excipients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 158 (Actual)
Dates: Start 2021-12-01 (Actual); Primary Completion 2024-03-06 (Actual); Study Completion 2024-03-06 (Actual)

PRIMARY OUTCOMES:
Positive predictive value (PPV) on a per-region- and per-patient-basis (table 3) of 68Ga-FAPI46 PET for detection of histopathology-FAP-positive tumor lesions, confirmed by histopathology/biopsy (reached for ≥ 75%). | within 8 weeks of FAPI-PET scan, when a tumor sample becomes available for immonostaining for FAP

SECONDARY OUTCOMES:
Correlation between 68Ga-FAPI-46 PET uptake intensity and histopathologic FAP expression | within 8 weeks of FAPI-PET scan, when a tumor sample becomes available for immonostaining for FAP
Sensitivity and specificity of FAPI-PET on a per-patient and per-region-basis for detection of histopathology-FAP-positive tumor lesions confirmed by histopathology/biopsy | within 8 weeks of FAPI-PET scan, when a tumor sample becomes available for immonostaining for FAP
Detection rate of FAPI-PET versus previous standard imaging on a per-patient and per-region-basis for detection of tumor location, also stratified by tumor maker serum level | up to time point when patient reaches end-of-study criterion (30day, if surgery is performed within 30 days after FAPI-PET or up to 8 weeks, at time of surgery/biopsy)
Sensitivity and specificity of FAPI-PET vs. previous standard imaging on a per-patient and per-region-basis for detection of tumor lesions confirmed by combined histo/biopsy/FU imaging/clinical FU reference standard | up to time point when patient reaches end-of-study criterion (30 day, if surgery is performed within 30 days after FAPI-PET or up to 8 weeks, at time of surgery/biopsy)
Inter-reader reproducibility: determination of FAPI-PET scan interpretation reliability by three independent evaluators | through study completion, an average of 1 year
Safety (AEs, SAEs, SUSARs) | From signing the ICF until day 30 after FAPI-PET scan
Change in staging/prognostic groups per survey of referring physician who was provided with FAPI-PET scan information. | through study completion, an average of 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Nuclear medicine, University hospital Essen, Essen, North Rhine-Westphalia, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pabst KM, Weber MM, Laschinsky C, Sandach P, Bartel T, Kuper AT, Kessler L, Trajkovic-Arsic M, Eckstein M, Gilman E, Nader M, Barbato F, Podleska LE, Hadaschik BA, Hamacher R, Kersting D, von Ostau N, von Tresckow B, Kaelberlah HP, Kesch C, Kuemmel S, Reinacher-Schick A, Schuler M, Siveke JT, Grunwald V, Herrmann K, Fendler WP. [68Ga]Ga-FAPI-46 PET accuracy for cancer imaging with histopathology validation: a single-centre, single-arm, interventional, phase 2 trial. Lancet Oncol. 2025 Sep;26(9):1204-1214. doi: 10.1016/S1470-2045(25)00299-2. Epub 2025 Aug 4. PMID 40774265
- [Derived] Watanabe M, Fendler WP, Grafe H, Hirmas N, Hamacher R, Lanzafame H, Pabst KM, Hautzel H, Aigner C, Kasper S, von Tresckow B, Stuschke M, Kummel S, Lugnier C, Hadaschik B, Grunwald V, Zarrad F, Kersting D, Siveke JT, Herrmann K, Weber M. Head-to-head comparison of 68 Ga-FAPI-46 PET/CT, 18F-FDG PET/CT, and contrast-enhanced CT for the detection of various tumors. Ann Nucl Med. 2025 Mar;39(3):255-265. doi: 10.1007/s12149-024-01993-7. Epub 2024 Oct 23. PMID 39443386
- [Derived] Hirmas N, Hamacher R, Sraieb M, Kessler L, Pabst KM, Barbato F, Lanzafame H, Kasper S, Nader M, Kesch C, von Tresckow B, Hautzel H, Aigner C, Glas M, Stuschke M, Kummel S, Harter P, Lugnier C, Uhl W, Hadaschik B, Grunwald V, Siveke JT, Herrmann K, Fendler WP. Diagnostic Accuracy of 68Ga-FAPI Versus 18F-FDG PET in Patients with Various Malignancies. J Nucl Med. 2024 Mar 1;65(3):372-378. doi: 10.2967/jnumed.123.266652. Epub 2024 Feb 8. PMID 38331453